CLINICAL TRIAL: NCT06474767
Title: Addressing Health Disparities in Chronic Lung Disease for Preterm Infants Through Parent Engagement
Brief Title: Using Parent Engagement to Improve the Wellbeing of Black Premature Infants With Chronic Lung Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00447949
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric Collaborative Goal Setting Participant (Experimental): Participants will receive pediatric collaborative goal setting (P-CGS) intervention one to three days prior to the child's identified well visit and will be asked to complete it before or at the time of the visit. Participants will identify 1 goal for the child's health and the parent's own health, covering both medical and social domains. Participants will then be prompted to share the content with the child's provider when asked about the parent's priorities during the child's visit. One week and two months after the child's well visit where pediatric collaborative goal setting was used, participants will complete follow up surveys.
  Interventions: Behavioral: P-CGS (Pediatric Collaborative Goal Setting)

INTERVENTIONS:
Behavioral: P-CGS (Pediatric Collaborative Goal Setting) — Electronic questionnaire sent to participants ahead of a pediatric primary care well child visit, assessing goals for themselves and the child's health with prompt to share with providers during visit

SUMMARY:
The goal of this pilot study is to test the feasibility and acceptability of a collaborative goal setting intervention to improve parent engagement of Black preterm infants with chronic lung disease in primary care. Preliminary impact on child and parent outcomes will also be explored.

The main questions it aims to answer are: 1) Will parents complete a pre-visit questionnaire that asks about goals for the child? 2) Does use of the pre-visit questionnaire help parents to achieve self-identified goals?

Participants will fill out a pre-visit questionnaire prior to the child's well visit. The participants will then complete two surveys after the visit (1 week and 2 months after).

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal guardian of child born prior to 37 weeks gestational age
* Parent/legal guardian of child with diagnosis of chronic lung disease or bronchopulmonary dysplasia, as defined by the child's clinical team at the time of hospital discharge
* Parent/legal guardian of child who identifies that child's race as Black
* English speaking

Exclusion Criteria:

* Parent/legal guardian of child enrolled in palliative care or hospice services at time of hospital discharge
* Parent/legal guardian of child older than 12 months chronological age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility as measured by number of interventions completed | Day 0
  Number of participants who complete the pediatric collaborative goal setting intervention out of the number of consented participants who are sent a link prior to the child's well visit
Feasibility as measured by the time it takes participant to complete intervention | Day 0
  Amount of time (minutes) that participant has the pediatric collaborative goal setting intervention open
Feasibility as measured by the number of goals submitted by each participant | Day 0
  Number of goals submitted by each participant through the pediatric collaborative goal setting intervention
Acceptability of the intervention as assessed by the Acceptability of Intervention Measure (AIM) scale | Day 7 post-intervention
  Measured by the Acceptability of Intervention Measure (AIM) scale - a 4 item survey with 5 point Likert scales from Completely Disagree to Completely Agree. Score ranges from 4 to 20, where higher scores indicate greater acceptability.

SECONDARY OUTCOMES:
Goal attainment as assessed by number of goals submitted | Day 60 post-intervention
  Number of goals submitted as part of pediatric collaborative goal setting that were accomplished by participant since intervention
Participation activation as measured by Parent Patient Activation Measure 10 | Day 60 post-intervention
  Measured by the Parent Patient Activation Measure scale - a 7 item survey with 4 point Likert scales (total score range 7-28) from Disagree Strongly to Agree Strongly with higher scores indicating a better outcome.
Participant's child's respiratory symptoms as measured by self-report | Day 60 post-intervention
  Frequency of rescue inhaler use and symptoms of wheezing, rated on 5 point Likert scale (total score range 1-5) from Never to Every day with higher scores indicating more use and worse outcome. This is a survey instrument constructed by the study team.
Participant's child's use of the emergency department for breathing symptoms as measured by self-report | Day 60 post-intervention
  Frequency of emergency department visits, rated on 5 point Likert scale (total score range 1-5) from Never to Every day with higher scores indicating more use and worse outcome. This is a survey instrument constructed by the study team.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon M Smith, MD MPH, Principal Investigator — Johns Hopkins School of Medicine